CLINICAL TRIAL: NCT04421027
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase 3 Study of Baricitinib in Patients With COVID-19 Infection
Brief Title: A Study of Baricitinib (LY3009104) in Participants With COVID-19
Acronym: COV-BARRIER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17830; I4V-MC-KHAA (Other: Eli Lilly and Company); 2020-001517-21 (EudraCT Number)
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Results first posted 2022-03-24 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: coronavirus; coronavirus infection; safety
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baricitinib + Standard of Care (SOC) (Experimental): 4 milligrams (mg) of baricitinib (given as two 2 mg tablets) administered orally every day (QD) with standard of care.
  Interventions: Drug: Baricitinib
- Placebo + SOC (Placebo Comparator): Placebo (given as two placebo tablets) administered orally QD with standard of care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Given orally
  Other Names: LY3009104
  Arms: Baricitinib + Standard of Care (SOC)
Drug: Placebo — Given orally
  Arms: Placebo + SOC

SUMMARY:
The reason for this study is to see if the study drug baricitinib is effective in hospitalized participants with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with coronavirus (SARS-CoV-2) infection, confirmed by polymerase chain reaction (PCR) test or other commercial or public health assay in any specimen, as documented by either of the following:

  * PCR positive in sample collected <72 hours prior to randomization; OR
  * PCR positive in sample collected ≥72 hours prior to randomization (but no more than 14 days prior to randomization), documented inability to obtain a repeat sample (for example, due to lack of testing supplies, limited testing capacity, results taking >24 hours, etc.) AND progressive disease suggestive of ongoing SARS-CoV-2 infection.
* Requires supplemental oxygen at the time of study entry and at randomization.
* Have indicators of risk of progression: at least 1 inflammatory markers >upper limit of normal (ULN) (C reactive protein [CRP], D dimer, lactate dehydrogenase [LDH], ferritin) with at least 1 instance of elevation >ULN within 2 days before study entry.

Exclusion Criteria:

* Are receiving cytotoxic or biologic treatments (such as tumor necrosis factor [TNF] inhibitors, anti-interleukin-1 [IL-1], anti-IL-6 [tocilizumab or sarilumab], T-cell or B-cell targeted therapies (rituximab), interferon, or Janus kinase (JAK) inhibitors for any indication at study entry. Note: A washout period 4 weeks (or 5 half-lives, whichever is longer) is required prior to screening.
* Have ever received convalescent plasma or intravenous immunoglobulin [IVIg]) for COVID-19.
* Have received high dose corticosteroids at doses >20 mg per day (or prednisone equivalent) administered for ≥14 consecutive days in the month prior to study entry.
* Strong inhibitors of OAT3 (such as probenecid) that cannot be discontinued at study entry.
* Have received neutralizing antibodies, such as bamlanivimab, casirivimab and imdevimab for COVID-19.
* Have diagnosis of current active tuberculosis (TB) or, if known, latent TB treated for less than 4 weeks with appropriate anti-tuberculosis therapy per local guidelines (by history only, no screening tests required).
* Suspected serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking investigational product.
* Have received any live vaccine within 4 weeks before screening, or intend to receive a live vaccine during the study. Note: Use of nonlive (inactivated) vaccinations is allowed for all participants.
* Require invasive mechanical ventilation, including extracorporeal membrane oxygenation (ECMO) at study entry.
* Current diagnosis of active malignancy that, in the opinion of the investigator, could constitute a risk when taking investigational product.
* Have a history of venous thromboembolism (VTE) (deep vein thrombosis [DVT] and/or pulmonary embolism [PE]) within 12 weeks prior to randomization or have a history of recurrent (>1) VTE (DVT/PE).
* Anticipated discharge from the hospital, or transfer to another hospital (or another unit), which is not a study site within 72 hours after study entry.
* Have neutropenia (absolute neutrophil count <1000 cells/microliters).
* Have lymphopenia (absolute lymphocyte count <200 cells/microliters).
* Have alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 times ULN.
* Estimated glomerular filtration rate (eGFR) (Modification of Diet in Renal Disease [MDRD]) <30 milliliter/minute/1.73 meters squared.
* Have a known hypersensitivity to baricitinib or any of its excipients.
* Are currently enrolled in any other clinical study involving an investigation product or any other type of medical research judged not to be scientifically or medically compatible with this study. Note: The participant should not be enrolled (started) in another clinical trial for the treatment of COVID-19 or SARS CoV-2 through Day 28.
* Are pregnant, or intend to become pregnant or breastfeed during the study.
* Are using or will use extracorporeal blood purification (EBP) device to remove proinflammatory cytokines from the blood such as a cytokine absorption or filtering device, for example, CytoSorb®.
* Are, in the opinion of the investigator, unlikely to survive for at least 48 hours after screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1525 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-265-4559 or 1-317-615-4559) Mon - Fri 9AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (96):
- United States (25):
  - Dignity Health Mercy Gilbert Medical Center, Gilbert, Arizona
  - Valleywise Health, Phoenix, Arizona
  - St Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Sharp Memorial Hospital, San Diego, California
  - San Francisco VA Medical Center, San Francisco, California
  - Torrance Memorial Medical Center, Torrance, California
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - Westchester General Hospital, Miami, Florida
  - Grady Health System, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Community Hospital South, Indianapolis, Indiana
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - South Shore Hospital, Weymouth, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Renown Regional Med. Center, Reno, Nevada
  - SUNY Downstate, Brooklyn, New York
  - East Carolina University, Greenville, North Carolina
  - OSU Med Intl Med Houston Ctr, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Temple Univ School of Med, Philadelphia, Pennsylvania
  - Swedish Medical Center, Seattle, Washington
  - MultiCare Good Samaritan Hospital, Tacoma, Washington
- Argentina (11):
  - Sanatorio Sagrado Corazón, Ciudad de Buenos Aires, AR
  - ClÃ-nica Zabala, Ciudad de Buenos Aires, AR
  - Hospital Z.G.A.D "Evita Pueblo", Berazategui, Buenos Aires
  - Sanatorio de la Trinidad Mitre, CABA, Buenos Aires
  - Fundacion Sanatorio Guemes, CABA, Buenos Aires
  - Casa Hospital San Juan de Dios, Ramos Mejía, Buenos Aires
  - Hospital Interzonal General de Agudos "Eva Peron", San Martín, Buenos Aires
  - Clinica Adventista Belgrano, CABA, Ciudad Autónoma de Buenos Aire
  - Clinica Viedma, Viedma, Río Negro Province
  - Clinica Central S.A., Villa Regina, Río Negro Province
  - Hospital San Roque, Córdoba
- Brazil (19):
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Centro Hospitalar de Reabilitacao Ana Carolina Moura Xavier, Curitiba, Paraná
  - CEPETI Centro de Ensino e Pesquisa em Terapia Intensiva, Curitiba, Paraná
  - CPCLIN, Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Upeclin - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu - UNESP, Botucatu, São Paulo
  - IPECC - Instituto de Pesquisa Clinica de Campinas, Campinas, São Paulo
  - Hospital PUC-CAMPINAS, Campinas, São Paulo
  - CECIP - Centro de Estudos do Interior Paulista, Jaú, São Paulo
  - Hospital Carlos Fernando Malzoni Matao, Matão, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Pesquisare, Santo André, São Paulo
  - Praxis Pesquisa Medica, Santo André, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clinicos EPP Ltda, São Bernardo do Campo, São Paulo
  - Real e Benemerita Associação Portuguesa de Beneficiencia, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - Universidade Federal de São Paulo - Escola Paulista de Medicina, São Paulo
  - Hospital Santa Paula, São Paulo
  - Casa de Saude Santa Marcelina - Centro de Pesquisa Clinica, São Paulo
- Germany (4):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum Rechts der Isar der TU München, München, Bavaria
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Klinikum Chemnitz gGmbH, Chemnitz
- India (8):
  - Unity Hospital, Surat, Gujarat
  - Medanta-The Medicity, Gurgaon, Haryana
  - Government Medical College (GMC) Aurangabad, Aurangabad, Maharashtra
  - Government Medical College, Nagpur, Maharashtra
  - Ruby Hall Clinic and Grant Medical Foundation, Pune, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Medica Superspecialty Hospital, Kolkata, West Bengal
  - Aakash Healthcare Super Speciality Hospital, New Delhi
- Italy (3):
  - INMI Lazzaro Spallanzani, Roma, Rome
  - Ospedale Niguarda Ca Granda, Milan
  - Nuovo Ospedale di Prato S. Stefano, Prato
- Japan (3):
  - Yokohama Municipal Citizen's Hospital, Yokohama, Kanagawa
  - Edogawa Medicare Hospital, Edagawa, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
- Mexico (7):
  - Instituto Nacional de Cancerologia, Mexico City, FD
  - Instituto Nacional de Ciencias Medicas y Nutrici Salva Zubir, Mexico City, Federal District
  - Hospital General Agustín O'Horán, Yucatán, Merida
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - ITESM Campus Monterrey, Monterrey, Nuevo León
- Advanced Clinical Research, LLC, Bayamón, PR, Puerto Rico
- Russia (3):
  - City Clinical Hospital #15 named after O.M. Filatov, Moscow
  - First Moscow State Medical University n.a. Sechenov, Moscow
  - Saint-Petersburg City Pokrovskaya Hospital, Saint Petersburg
- South Korea (4):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Seoul National University Boramae Medical Center, Seoul, Seoul, Korea
  - Seoul Medical Center, Seoul
- Spain (5):
  - Hospital Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Infanta Leonor-INTERNAL MED, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (3):
  - The Royal Cornwall Hospital, Truro, Cornwall
  - Barnet Hospital, Barnet, Herts
  - St. George's University Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting
Access Criteria: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting
URL: http://vivli.org/

REFERENCES:
- [Derived] Kramer A, Prinz C, Fichtner F, Fischer AL, Thieme V, Grundeis F, Spagl M, Seeber C, Piechotta V, Metzendorf MI, Golinski M, Moerer O, Stephani C, Mikolajewska A, Kluge S, Stegemann M, Laudi S, Skoetz N. Janus kinase inhibitors for the treatment of COVID-19. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD015209. doi: 10.1002/14651858.CD015209. PMID 35695334
- [Derived] Ely EW, Ramanan AV, Kartman CE, de Bono S, Liao R, Piruzeli MLB, Goldman JD, Saraiva JFK, Chakladar S, Marconi VC; COV-BARRIER Study Group. Efficacy and safety of baricitinib plus standard of care for the treatment of critically ill hospitalised adults with COVID-19 on invasive mechanical ventilation or extracorporeal membrane oxygenation: an exploratory, randomised, placebo-controlled trial. Lancet Respir Med. 2022 Apr;10(4):327-336. doi: 10.1016/S2213-2600(22)00006-6. Epub 2022 Feb 3. PMID 35123660
- [Derived] Marconi VC, Ramanan AV, de Bono S, Kartman CE, Krishnan V, Liao R, Piruzeli MLB, Goldman JD, Alatorre-Alexander J, de Cassia Pellegrini R, Estrada V, Som M, Cardoso A, Chakladar S, Crowe B, Reis P, Zhang X, Adams DH, Ely EW; COV-BARRIER Study Group. Efficacy and safety of baricitinib for the treatment of hospitalised adults with COVID-19 (COV-BARRIER): a randomised, double-blind, parallel-group, placebo-controlled phase 3 trial. Lancet Respir Med. 2021 Dec;9(12):1407-1418. doi: 10.1016/S2213-2600(21)00331-3. Epub 2021 Sep 1. PMID 34480861
- See also: A Study of Baricitinib (LY3009104) in Participants With COVID-19 (COV-BARRIER) — https://trials.lillytrialguide.com/en-US/trial/1QT4STirLDGakzCVTBX2Rv

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Standard of Care (SOC): Placebo tablets administered orally every day (QD) with standard of care.
- Baricitinib + SOC: 4 milligrams (mg) baricitinib administered orally QD with standard of care.
- Placebo + SOC Follow-Up; Baricitinib + SOC Follow-Up: Participants did not receive drug during the Follow-Up Period.
Period: Treatment Period
Arm/Group | Placebo + Standard of Care (SOC) | Baricitinib + SOC | Placebo + SOC Follow-Up | Baricitinib + SOC Follow-Up
Started | 761 | 764 | 0 | 0
Received at Least One Dose of Study Drug | 752 | 750 | 0 | 0
Completed | 604 | 644 | 0 | 0
Not Completed | 157 | 120 | 0 | 0
Not completed — Adverse Event | 5 | 3 | 0 | 0
Not completed — Death | 98 | 61 | 0 | 0
Not completed — Lost to Follow-up | 22 | 20 | 0 | 0
Not completed — Other-Unknown | 15 | 9 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 12 | 0 | 0
Not completed — Randomized Not Dosed | 9 | 14 | 0 | 0
Period: Follow-Up Period
Arm/Group | Placebo + Standard of Care (SOC) | Baricitinib + SOC | Placebo + SOC Follow-Up | Baricitinib + SOC Follow-Up
Started | 0 | 0 | 613 | 645
Completed | 0 | 0 | 588 | 615 (One participants study disposition case report form was not completed, therefore the participant appeared as 'ongoing' at Day 60. The participant completed Day 60 Clinical Status Assessment (CSA) and is considered as completing the study.)
Not Completed | 0 | 0 | 25 | 30
Not completed — Adverse Event | 0 | 0 | 0 | 3
Not completed — Death | 0 | 0 | 16 | 17
Not completed — Lost to Follow-up | 0 | 0 | 7 | 7
Not completed — Protocol Deviation | 0 | 0 | 1 | 0
Not completed — Still in hospital on ventilator at end of study | 0 | 0 | 1 | 0
Not completed — Left message, participant did not call back | 0 | 0 | 0 | 1
Not completed — Participant died | 0 | 0 | 0 | 1
Not completed — Participant was alive but did not respond to calls | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants randomly assigned to study intervention. Participants were analyzed according to the intervention to which they were assigned.
Groups:
- Placebo +SOC: Placebo administered orally QD with standard of care.
- Baricitinib + SOC: 4 mg baricitinib administered orally QD with standard of care.
- Total: Total of all reporting groups
Arm/Group | Placebo +SOC | Baricitinib + SOC | Total
Number analyzed (Participants) | 761 | 764 | 1525
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (13.8) | 57.8 (14.3) | 57.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 288 | 274 | 562
  Male | 473 | 490 | 963
Race (NIH/OMB) [Count of Participants; unit: Participants] — American Indian or Alaska Native category includes participants from Mexico and Latin America.
  Participants
    American Indian or Alaska Native | 168 | 148 | 316
    Asian | 94 | 80 | 174
    Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
    Black or African American | 36 | 39 | 75
    White | 440 | 480 | 920
    More than one race | 1 | 2 | 3
    Unknown or Not Reported | 20 | 12 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 3 | 8 | 11
  Argentina | 101 | 107 | 208
  United States | 155 | 154 | 309
  Japan | 19 | 19 | 38
  United Kingdom | 7 | 4 | 11
  India | 31 | 19 | 50
  Russia | 54 | 58 | 112
  Spain | 42 | 45 | 87
  South Korea | 20 | 16 | 36
  Brazil | 165 | 172 | 337
  Mexico | 143 | 138 | 281
  Italy | 10 | 15 | 25
  Germany | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Die or Require Non-Invasive Ventilation/High-Flow Oxygen or Invasive Mechanical Ventilation (Including Extracorporeal Membrane Oxygenation [ECMO])
Description: Percentage of participants who die or require non-invasive ventilation/high-flow oxygen or invasive mechanical ventilation (including ECMO).
Time Frame: Day 1 to Day 28
Population: All participants randomly assigned to study intervention. Participants with missing baseline ordinal scale values were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo + SOC: Placebo administered orally QD with standard of care.
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 756 | 762
percentage of participants | 30.5 [27.2 to 33.8] | 27.8 [24.6 to 31.0]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.1800, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.67 to 1.08]

2. Primary Outcome: Percentage of Participants Who Die or Require Non-Invasive Ventilation/High-Flow Oxygen or Invasive Mechanical Ventilation (Including Extracorporeal Membrane Oxygenation [ECMO] Population 2
Description: Percentage of participants who die or require non-invasive ventilation or invasive mechanical ventilation, including ECMO.
Time Frame: Day 1 to Day 28
Population: All participants randomly assigned to study intervention who at baseline required oxygen supplementation and did not receive dexamethasone, or other systemic corticosteroids for the primary study condition.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 109 | 96
percentage of participants | 27.1 [18.7 to 35.6] | 28.9 [19.6 to 38.2]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.7280, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.58 to 2.16]

3. Secondary Outcome: Percentage of Participants With at Least 1-Point Improvement on National Institute of Allergy and Infectious Diseases Ordinal Scale (NIAID-OS) or Live Discharge From Hospital
Description: The National Institute of Allergy and Infectious Diseases ordinal scale (NIAID-OS) is an assessment of clinical status. The scale is as follows: 1) Not hospitalized, no limitations on activities; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 5) Hospitalized, requiring supplemental oxygen; 6) Hospitalized, on non-invasive ventilation or high-flow oxygen devices; 7) Hospitalized, on invasive mechanical ventilation or ECMO; 8) Death. Participants with missing baseline ordinal scale values were excluded from analysis.
Time Frame: Day 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 756 | 762
percentage of participants | 63.5 [60.1 to 67.0] | 65.0 [61.6 to 68.5]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.5444, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.86 to 1.34]

4. Secondary Outcome: Number of Ventilator-Free Days
Description: Number of days free of invasive mechanical ventilation.
Time Frame: Day 1 to Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 756 | 762
days | 23.7 (0.39) | 24.5 (0.39)
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.0586, ANOVA; LS Mean difference (net) = 0.75, 95% CI 2-sided [-0.0 to 1.5], Standard Error of Mean 0.399

5. Secondary Outcome: Time to Recovery
Description: Recovery assessed by the National Institute of Allergy and Infectious Diseases Ordinal Scale (NIAID-OS). Time to reach NIAID-OS 1, 2, or 3 for the first time. The date reached is the first full day that OS 1, 2, or 3 is the participant's maximum OS for the day.
  NIAID-OS 1. Not hospitalized, no limitations on activities 2. Not hospitalized, limitation on activities and/or requiring home oxygen 3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care: (This would include those kept in hospital for quarantine/infection control, awaiting bed in rehabilitation facility or homecare, etc.)
Time Frame: Day 1 to Day 28
Population: All participants randomly assigned to study intervention.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 761 | 764
days | 11.0 [10.0 to 12.0] | 10.0 [9.0 to 11.0]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.1453, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.99 to 1.24]

6. Secondary Outcome: Percentage of Participants at Each Clinical Status Using the National Institute of Allergy and Infectious Diseases Ordinal Scale (NIAID-OS) at Day 4
Description: Overall improvement on the National Institute of Allergy and Infectious Diseases ordinal scale:
  1. Not hospitalized, no limitations on activities; 2. Not hospitalized, limitation on activities and/or requiring home oxygen; 3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care: (This would include those kept in hospital for quarantine/infection control, awaiting bed in rehabilitation facility or homecare, etc.); 4. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 5. Hospitalized, requiring supplemental oxygen; 6.Hospitalized, on noninvasive ventilation or high-flow oxygen devices; 7. Hospitalized, on invasive mechanical ventilation or ECMO; 8. Death.
Time Frame: Day 4
Population: All participants randomly assigned to study intervention. Participants with missing baseline ordinal scale were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 756 | 762
percentage of participants
  Day 4 NIAID-OS 1 | 4.6 [3.1 to 6.1] | 5.2 [3.6 to 6.8]
  Day 4 NIAID-OS 2 | 1.5 [0.6 to 2.4] | 1.5 [0.6 to 2.4]
  Day 4 NIAID-OS 3 | 0.8 [0.2 to 1.4] | 0.3 [0.0 to 0.7]
  Day 4 NIAID-OS 4 | 19.4 [16.6 to 22.3] | 23.6 [20.6 to 26.7]
  Day 4 NIAID-OS 5 | 41.0 [37.5 to 44.5] | 39.0 [35.5 to 42.5]
  Day 4 NIAID-OS 6 | 22.4 [19.5 to 25.4] | 21.8 [18.9 to 24.8]
  Day 4 NIAID-OS 7 | 8.9 [6.8 to 10.9] | 8.1 [6.2 to 10.1]
  Day 4 NIAID-OS 8 | 1.4 [0.5 to 2.2] | 0.4 [0.0 to 0.9]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Day 4; Test type: Superiority; p = 0.0464, Proportional Odds Model; Odds Ratio (OR) = 1.21, 95% CI 2-sided [1.00 to 1.47]

7. Secondary Outcome: Percentage of Participants at Each Clinical Status Using the National Institute of Allergy and Infectious Diseases Ordinal Scale (NIAID-OS) at Day 7
Description: as for outcome 6
Time Frame: Day 7
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 756 | 762
percentage of participants
  Day 7 NIAID-OS 1 | 20.2 [17.3 to 23.1] | 25.2 [22.1 to 28.4]
  Day 7 NIAID-OS 2 | 6.6 [4.8 to 8.4] | 5.8 [4.1 to 7.5]
  Day 7 NIAID-OS 3 | 0.5 [0.0 to 1.1] | 0.2 [0.0 to 0.5]
  Day 7 NIAID-OS 4 | 21.2 [18.2 to 24.1] | 20.6 [17.6 to 23.5]
  Day 7 NIAID-OS 5 | 22.5 [19.5 to 25.5] | 22.5 [19.4 to 25.5]
  Day 7 NIAID-OS 6 | 14.5 [12.0 to 17.0] | 13.8 [11.3 to 16.2]
  Day 7 NIAID-OS 7 | 11.2 [9.0 to 13.5] | 10.8 [8.6 to 13.0]
  Day 7 NIAID-OS 8 | 3.3 [2.0 to 4.5] | 1.2 [0.4 to 2.0]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.0172, Proportional Odds Model; Odds Ratio (OR) = 1.25, 95% CI 2-sided [1.04 to 1.49]

8. Secondary Outcome: Percentage of Participants at Each Clinical Status Using the National Institute of Allergy and Infectious Diseases Ordinal Scale (NIAID-OS) at Day 10
Description: as for outcome 6
Time Frame: Day 10
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 756 | 762
percentage of participants
  Day 10 NIAID-OS 1 | 37.7 [34.2 to 41.2] | 40.4 [36.9 to 44.0]
  Day 10 NIAID-OS 2 | 9.4 [7.3 to 11.5] | 10.9 [8.7 to 13.2]
  Day 10 NIAID-OS 3 | 0.1 [0.0 to 0.4] | 0.1 [0.0 to 0.4]
  Day 10 NIAID-OS 4 | 16.2 [13.6 to 18.9] | 14.1 [11.6 to 16.6]
  Day 10 NIAID-OS 5 | 12.8 [10.3 to 15.2] | 12.4 [10.0 to 14.8]
  Day 10 NIAID-OS 6 | 8.1 [6.1 to 10.0] | 8.9 [6.8 to 11.0]
  Day 10 NIAID-OS 7 | 10.6 [8.4 to 12.9] | 10.4 [8.2 to 12.6]
  Day 10 NIAID-OS 8 | 5.1 [3.5 to 6.7] | 2.6 [1.5 to 3.8]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.0921, Proportional Odds Model; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.97 to 1.41]

9. Secondary Outcome: Percentage of Participants at Each Clinical Status Using the National Institute of Allergy and Infectious Diseases Ordinal Scale (NIAID-OS) at Day 14
Description: as for outcome 6
Time Frame: Day 14
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 756 | 762
percentage of participants
  Day 14 NIAID-OS 1 | 51.6 [48.0 to 55.2] | 56.3 [52.7 to 59.9]
  Day 14 NIAID-OS 2 | 11.2 [8.9 to 13.5] | 11.1 [8.8 to 13.4]
  Day 14 NIAID-OS 3 | 0.3 [0.0 to 0.6] | 0.1 [0.0 to 0.4]
  Day 14 NIAID-OS 4 | 8.0 [6.0 to 10.0] | 7.6 [5.7 to 9.6]
  Day 14 NIAID-OS 5 | 8.4 [6.4 to 10.5] | 7.3 [5.4 to 9.2]
  Day 14 NIAID-OS 6 | 3.6 [2.2 to 4.9] | 3.7 [2.3 to 5.1]
  Day 14 NIAID-OS 7 | 9.4 [7.3 to 11.6] | 8.9 [6.9 to 11.0]
  Day 14 NIAID-OS 8 | 7.5 [5.6 to 9.4] | 4.9 [3.4 to 6.5]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.0168, Proportional Odds Model; Odds Ratio (OR) = 1.28, 95% CI 2-sided [1.05 to 1.56]

10. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization.
Time Frame: Days 1 to Day 28
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 756 | 762
days | 13.7 (0.40) | 12.9 (0.40)
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.0626, ANOVA; LS Mean Difference (Net) = -0.76, 95% CI 2-sided [-1.6 to 0.0], Standard Error of Mean 0.408

11. Secondary Outcome: Percentage of Participants With a Change in Oxygen Saturation From < 94% to ≥ 94% From Baseline
Description: Percentage of participants with a change in oxygen saturation from < 94% to ≥ 94% from baseline based on National Early Warning Score (NEWS). Measure of the oxygen level of the blood is measure by pulse oximetry. The score is determined from six physiological parameters readily measured over time in hospitalized participants: Respiration rate; oxygen saturation; temperature; systolic blood pressure; heart (pulse) rate, and level of consciousness, as measured by Alert Voice Pain Unresponsive (AVPU). A score is assigned to each parameter, the magnitude of the score representing the extremity of variation from the norm. A weighting score is added for participants needing supplemental oxygen (oxygen delivery by mask or by cannula) The aggregate score is reflective of the participants status.
Time Frame: Day 10
Population: All participants randomly assigned to study intervention whose oxygen saturation (based on National Early Warning Score) is < 94% at baseline and have non-missing baseline and at least 1 postbaseline observation are in this population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 282 | 282
percentage of participants | 52.5 [46.7 to 58.2] | 56.7 [50.9 to 62.4]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.4290, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.81 to 1.63]

12. Secondary Outcome: Overall Mortality
Description: Number of deaths by Day 28.
Time Frame: Day 1 to Day 28
Population: All participants randomly assigned to study intervention.
Measure: Number; unit: event of death
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 761 | 764
event of death | 104 | 65
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.0018, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.41 to 0.78]

13. Secondary Outcome: Duration of Stay in the Intensive Care Unit (ICU) in Days
Description: Duration of stay in the ICU in days.
Time Frame: Day 1 to Day 28
Population: All participants randomly assigned to study intervention with non-missing baseline NIAID OS and at least 1 postbaseline NIAID OS observation.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 754 | 758
days | 3.17 (0.313) | 3.19 (0.315)
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.9526, ANOVA; LS Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.62 to 0.65], Standard Error of Mean 0.323

14. Secondary Outcome: Time to Clinical Deterioration (One-category Increase on the NIAID-OS)
Description: The National Institute of Allergy and Infectious Diseases ordinal scale (NIAID-OS) is an assessment of clinical status. The scale is as follows: 1) Not hospitalized, no limitations on activities; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 5) Hospitalized, requiring supplemental oxygen; 6) Hospitalized, on non-invasive ventilation or high-flow oxygen devices; 7) Hospitalized, on invasive mechanical ventilation or ECMO; 8) Death. A higher score is representative of worse clinical outcome with a score of 8 being the highest and representing death.
Time Frame: Day 1 to Day 28
Population: All participants randomly assigned to study intervention. Participants with missing baseline ordinal scale values were excluded from analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 761 | 764
days | NA [NA to NA] — Median not evaluable due to less than half the participants meeting criteria. | NA [NA to NA] — Median not evaluable due to less than half the participants meeting criteria.
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.1831, Log Rank; Hazard Ratio (HR) = 0.887, 95% CI 2-sided [0.741 to 1.061]

15. Secondary Outcome: Time to Resolution of Fever in Participants With Fever at Baseline
Description: Time to resolution of fever in participants with fever at baseline was calculated using cox proportional hazard regression model adjusted for baseline disease severity (OS 4, OS 5, OS 6), age (<65 years, >=65 years), region (United States, Europe, rest of world), and systemic corticosteroids used at baseline for primary study condition (Yes/No).
Time Frame: Day 1 to Day 28
Population: All participants randomly assigned to study intervention who had a fever at baseline.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 354 | 357
days | 4.00 [3.00 to 4.00] | 3.00 [3.00 to 4.00]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.0243, Log Rank; Hazard Ratio (HR) = 1.202, 95% CI 2-sided [1.017 to 1.421]

16. Secondary Outcome: Mean Change From Baseline on the National Early Warning Score (NEWS)
Description: The NEWS score is used to detect and report changes in illness severity in participants with acute illness to identify participants at risk for poor outcomes. The score is based on six physiological parameters (Respiration rate; oxygen saturation; temperature; systolic blood pressure; heart (pulse) rate, and level of consciousness). A score is assigned to each parameter, and the sum of the score represents the participant's risk of poor outcomes with a minimum score of 0 representing the better outcome, a score of 7 or greater reflects high clinical risk for worsening and maximum score of 19 representing the worse outcome.
Time Frame: Baseline, Day 4; Baseline, Day 7; Baseline, Day 10; Baseline, Day 14
Population: All participants randomly assigned to study intervention with baseline and 1 postbaseline observation.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 636 | 647
score on a scale
  Day 4 | -0.59 (0.127) | -0.76 (0.125)
  Day 7: number analyzed (Participants) | 488 | 485
  Day 7 | -0.86 (0.145) | -1.04 (0.143)
  Day 10: number analyzed (Participants) | 388 | 399
  Day 10 | -1.33 (0.160) | -1.45 (0.158)
  Day 14: number analyzed (Participants) | 300 | 299
  Day 14 | -1.41 (0.183) | -1.66 (0.182)
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Day 4; Test type: Superiority; p = 0.191, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.42 to 0.08], Standard Error of Mean 0.128
Statistical Analysis 2: Comparison: Placebo + SOC vs Baricitinib + SOC; Day 7; Test type: Superiority; p = 0.278, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.49 to 0.14], Standard Error of Mean 0.161
Statistical Analysis 3: Comparison: Placebo + SOC vs Baricitinib + SOC; Day 10; Test type: Superiority; p = 0.496, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.49 to 0.24], Standard Error of Mean 0.187
Statistical Analysis 4: Comparison: Placebo + SOC vs Baricitinib + SOC; Day 14; Test type: Superiority; p = 0.263, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.70 to 0.19], Standard Error of Mean 0.226

17. Secondary Outcome: Time to Definitive Extubation
Description: Time to definitive extubation included participants who progressed to OS 7 at any time prior to Day 28.
Time Frame: Day 1 to Day 28
Population: All participants randomly assigned to study intervention who were intubated at some point during the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 136 | 125
days | NA [NA to NA] — Median not evaluable due to less than half the participants meeting criteria. | NA [NA to NA] — Median not evaluable due to less than half the participants meeting criteria.

18. Secondary Outcome: Time to Independence From Non-Invasive Mechanical Ventilation
Description: Time to independence from non-invasive mechanical ventilation was measured in days among participants who required non-invasive ventilation.
Time Frame: Day 1 to Day 28
Population: All participants randomly assigned to study intervention whose baseline OS was 6 and were on non-invasive mechanical ventilation.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 187 | 183
days | 11.00 [9.00 to 13.00] | 12.00 [9.00 to 14.00]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.6436, Log Rank; Hazard Ratio (HR) = 1.090

19. Secondary Outcome: Time to Independence From Oxygen Therapy in Days
Description: Time to independence from oxygen therapy in days.
Time Frame: Day 1 to Day 28
Population: All randomized participants who had an ordinal scale score of 5 or 6 at baseline.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 659 | 673
days | 8.00 [8.00 to 9.00] | 8.00 [7.00 to 8.00]
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.1270, Log Rank; Hazard Ratio (HR) = 1.124

20. Secondary Outcome: Number of Days With Supplemental Oxygen Use
Description: Number of days with supplemental oxygen use.
Time Frame: Day 1 to Day 28
Population: All participants randomly assigned to study intervention who have non-missing baseline and at least 1 postbaseline observation.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 754 | 758
days | 4.60 (0.221) | 4.37 (0.222)
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.3058, ANOVA; LS Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.68 to 0.21], Standard Error of Mean 0.228

21. Secondary Outcome: Number of Days of Resting Respiratory Rate <24 Breaths Per Minute
Description: Number of days of resting respiratory rate <24 breaths per minute.
Time Frame: Day 1 to Day 28
Population: All participants randomly assigned to study intervention who had non-missing baseline and at least 1 postbaseline respiratory rate.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo + SOC | Baricitinib + SOC
Number analyzed (Participants) | 743 | 745
days | 9.62 (0.300) | 9.73 (0.304)
Statistical Analysis 1: Comparison: Placebo + SOC vs Baricitinib + SOC; Test type: Superiority; p = 0.7073, ANOVA; LS Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.49 to 0.72], Standard Error of Mean 0.306

ADVERSE EVENTS:
Time Frame: Baseline up to 119 days Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Description: All randomized participants who received at least 1 dose of study drug including participants who entered the post-treatment follow-up (f/u) period. The main study period included all events from the start of first dose to 28 days post dose. One participant receiving baricitinib had 2 events with fatal outcomes. One event occurred in the main study period and the second event occurred in the f/u period which resulted in the participant death being counted in both the main study and f/u periods.
Groups:
- Placebo: Placebo tablets administered orally every day (QD) with standard of care.
- 4 Milligrams (mg) Baricitinib: 4 milligrams (mg) baricitinib administered orally QD with standard of care.
- Placebo Follow-up; 4mg Baricitinib Follow-up: Participants did not receive drug during the Follow-Up Period.
Arm/Group | Placebo | 4 Milligrams (mg) Baricitinib | Placebo Follow-up | 4mg Baricitinib Follow-up
All-Cause Mortality (participants affected / at risk) | 104/752 | 65/750 | 16/613 | 18/645
Serious Adverse Events (participants affected / at risk) | 135/752 | 110/750 | 12/613 | 18/645
Other Adverse Events (participants affected / at risk) | 0/752 | 0/750 | 0/613 | 0/645
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=752) | 4 Milligrams (mg) Baricitinib (N=750) | Placebo Follow-up (N=613) | 4mg Baricitinib Follow-up (N=645)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 6 (6) | 3 (3) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 5 (5) | 4 (4) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 10 (10) | 8 (8) | 1 (1) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 21 (21) | 21 (21) | 0 (0) | 0 (0)
Device related bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 8 (8) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 4 (5) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 24 (24) | 13 (13) | 4 (4) | 5 (5)
Severe acute respiratory syndrome (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Fibrin d dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 10 (10) | 7 (7) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 0/473 (0) | 0/490 (0) | 1/377 (1) | 0/415 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 29 (29) | 17 (17) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 12 (12) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 10 (10) | 0 (0) | 1 (1)
Palliative care (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT04421027/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT04421027/SAP_001.pdf